CLINICAL TRIAL: NCT05387304
Title: A Follow-up Study of Asymptomatic Infections and Diagnosed Patients With Covid-19 in Shanghai
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCAM2022-1
Record Dates: First submitted 2022-05-23; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 infections: SARS-Cov-2 RNA postive

SUMMARY:
This study is to clarify the distribution characteristics, host and clinical characteristics, disease outcome and risk factors, changes of multiple organs such as cardiopulmonary function and changes in social and psychological indicators during long-term follow-up of omicron variant asymptomatic infections and diagnosed patients

ELIGIBILITY:
Inclusion Criteria:

* SARS-Cov-2-RNA positive
* informed consent signed

Exclusion Criteria:

* informed consent rejected

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: asymptomatic infections and diagnosed patients with COVID-19 in fangcang shelter hospitals in Shanghai
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
long-term outcomes，changes of clinical characteristic and social psychology | 10 years
  the 3rd，6th，9th month，average one year discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, Ph D, Principal Investigator — Ruijin Hospital; Erzhen Chen, Ph D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The data are not publicity available due to privacy and ethical restrictions